CLINICAL TRIAL: NCT02892500
Title: Single-site, Double Blinded, Randomized Investigation of Corticosteroid Versus Placebo Injection Under Ultrasound Guidance in Patients With Syndesmotic Ligament Injury or High Ankle Sprain
Brief Title: Investigation of Corticosteroid Versus Placebo Injection in Patients With Syndesmotic Ligament Injury or High Ankle Sprain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to enroll subjects
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SanfordHealth
Record Dates: First submitted 2016-08-23; First posted 2016-09-08 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries | interventions — Bupivacaine; betamethasone sodium phosphate; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine hydrochloride and betamethasone sodium phosphate (Experimental): When the patient has been randomized to either group, a licensed provider under the direction of the PI, will utilize the ultrasound to identify the inferior tibiofibular ligament (syndesmotic ligament). This provider that performs the injection will not be involved in any follow-up visits or return to play review. When appropriate positioning is confirmed the area will be injected with a mixture of 5 ml of 0.25 % bupivacaine hydrochloride and 2 ml of 3 mg/ml betamethasone sodium phosphate (Celestone® Soluspan®) (BTM)
  Interventions: Drug: bupivacaine hydrochloride and betamethasone sodium phosphate
- bupivacaine hydrochloride (Active Comparator): When the patient has been randomized to either group, a licensed provider under the direction of the PI, will utilize the ultrasound to identify the inferior tibiofibular ligament (syndesmotic ligament). This provider that performs the injection will not be involved in any follow-up visits or return to play review. When appropriate positioning is confirmed, the area will be injected with 5ml of bupivacaine hydrochloride.
  Interventions: Drug: bupivacaine hydrochloride

INTERVENTIONS:
Drug: bupivacaine hydrochloride and betamethasone sodium phosphate — 5ml of 0.25% bupivacaine hydrochloride and 2 ml of 3mg/ml betamethasone sodium phosphate one injection into the inferior tibiofibular ligament
  Other Names: Marcaine, Celestone, Soluspan,
  Arms: bupivacaine hydrochloride and betamethasone sodium phosphate
Drug: bupivacaine hydrochloride — 5ml of bupivacaine hydrochloride into the tibiofibular ligament
  Other Names: Marcaine
  Arms: bupivacaine hydrochloride

SUMMARY:
This study evaluates the use of corticosteroids acutely as an adjuvant treatment of the high ankle sprain. Subjects will receive either a corticosteroid or a local anesthetic injection.

DETAILED DESCRIPTION:
The term "high ankle sprain" refers to injury to the syndesmotic ligaments of the ankle. It has become a much more common injury comprising up to 24.6% of all ankle sprains , with an incidence of 2.4 per 1000 athlete exposures. These can present a significant therapeutic challenge for the sports physician and typically result in a prolonged morbidity and delayed return to activity. The literature shows a lack of information for definitive care of these athletes. Typical recovery for the high ankle sprain is almost twice as long as the more common lateral ankle inversion sprain with a mean time to return to play of 45 days. There is also a higher incidence of residual chronic pain comparing high ankle sprains to an isolated lateral ankle sprain. The current standard for treatment of this injury has been to depend on symptomatic treatment with an initial phase of rest and protected splinting. This is followed by the use of NSAID's with a graduated rehabilitation program to reduce swelling, improve range of motion, and regain strength and proprioception of the ankle. This is followed by protective taping or bracing and return to activities as tolerated. Inflammation is one of the body's first reactions to injury. Release of damaged cells and tissue debris occurs upon injury. These expelled particles act as antigens to stimulate a nonspecific immune response and to cause the proliferation of leukocytes. Local blood flow increases to transport the polymorphonuclear leukocytes, macrophages, and plasma proteins to the injured area. A redistribution of arteriolar flow produces stasis and hypoxia at the injury site. The resulting infiltration of tissues by the leukocytes, plasma proteins, and fluid causes the redness, swelling, and pain that are characteristic of inflammation. Initially, the inflammatory reaction serves several important purposes. The influx of leukocytes facilitates the process of phagocytosis and the removal of damaged cells and other particulate matter. Pain and tenderness remind the patient to protect the injured area; however, the inflammatory reaction eventually becomes counterproductive. The mechanism of corticosteroid action includes a reduction of the inflammatory reaction by limiting the capillary dilatation and permeability of the vascular structures. These compounds restrict the accumulation of polymorphonuclear leukocytes and macrophages and reduce the release of vasoactive kinins. They also inhibit the release of destructive enzymes that attack the injury debris and destroy normal tissue indiscriminately. Additionally, new research suggests that corticosteroids may inhibit the release of arachidonic acid from phospholipids, thereby reducing the formation of prostaglandins, which contribute to the inflammatory process. There are no previous prospective, randomized studies that look at utilization of corticosteroids in treatment of the high ankle sprain. Only anecdotal information is available in simple case reports for treatment. There was one study looking at treatment with platelet rich plasma injection which demonstrated shorter return to play times and less long term residual pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Musculoskeletal ultrasound performed which demonstrates injury pattern consistent with high ankle sprain.
* Must sign the informed consent form and agree to meet the needs of the study
* Clinically and ultra sound confirmed and isolated syndesmotic ligament injury or high ankle sprain without associated fracture
* Injury occurred within the previous 7 days

Exclusion Criteria:

* Surgical intervention required to stabilize the ankle
* Unable to read and understand the consent form
* Unable to meet the needs of the follow-up examinations
* Allergic to the betamethasone
* Current fungal infection
* Pregnancy or currently breast feeding

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Piatt, MD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- Sanford Orthopedics and Sports Medicine, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hunt KJ, George E, Harris AH, Dragoo JL. Epidemiology of syndesmosis injuries in intercollegiate football: incidence and risk factors from National Collegiate Athletic Association injury surveillance system data from 2004-2005 to 2008-2009. Clin J Sport Med. 2013 Jul;23(4):278-82. doi: 10.1097/JSM.0b013e31827ee829. PMID 23339895
- [Background] Hopkinson WJ, St Pierre P, Ryan JB, Wheeler JH. Syndesmosis sprains of the ankle. Foot Ankle. 1990 Jun;10(6):325-30. doi: 10.1177/107110079001000607. PMID 2113510
- [Background] Wright RW, Barile RJ, Surprenant DA, Matava MJ. Ankle syndesmosis sprains in national hockey league players. Am J Sports Med. 2004 Dec;32(8):1941-5. doi: 10.1177/0363546504264581. PMID 15572325
- [Background] Katznelson A, Lin E, Militiano J. Ruptures of the ligaments about the tibio-fibular syndesmosis. Injury. 1983 Nov;15(3):170-2. doi: 10.1016/0020-1383(83)90007-4. PMID 6642626
- [Background] Nussbaum ED, Hosea TM, Sieler SD, Incremona BR, Kessler DE. Prospective evaluation of syndesmotic ankle sprains without diastasis. Am J Sports Med. 2001 Jan-Feb;29(1):31-5. doi: 10.1177/03635465010290011001. PMID 11206253
- [Background] Cole BJ, Schumacher HR Jr. Injectable corticosteroids in modern practice. J Am Acad Orthop Surg. 2005 Jan-Feb;13(1):37-46. doi: 10.5435/00124635-200501000-00006. PMID 15712981
- [Background] Mei-Dan O, Kots E, Barchilon V, Massarwe S, Nyska M, Mann G. A dynamic ultrasound examination for the diagnosis of ankle syndesmotic injury in professional athletes: a preliminary study. Am J Sports Med. 2009 May;37(5):1009-16. doi: 10.1177/0363546508331202. Epub 2009 Mar 31. PMID 19336613
- [Background] Laver L, Carmont MR, McConkey MO, Palmanovich E, Yaacobi E, Mann G, Nyska M, Kots E, Mei-Dan O. Plasma rich in growth factors (PRGF) as a treatment for high ankle sprain in elite athletes: a randomized control trial. Knee Surg Sports Traumatol Arthrosc. 2015 Nov;23(11):3383-92. doi: 10.1007/s00167-014-3119-x. Epub 2014 Jun 18. PMID 24938396

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were randomized or treated during the study.
Period: Overall Study
Arm/Group | Bupivacaine Hydrochloride and Betamethasone Sodium Phosphate | Bupivacaine Hydrochloride
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized or treated therefore no baseline characteristics were collected for this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Hydrochloride and Betamethasone Sodium Phosphate | Bupivacaine Hydrochloride | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Compare Between the Two Groups the Time to Return to Previous Levels of Activity
Time Frame: One year
Population: No participants randomized and treated.
Arm/Group | Bupivacaine Hydrochloride and Betamethasone Sodium Phosphate | Bupivacaine Hydrochloride
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare Patient Reported Outcomes Between the Two Groups Using the Foot and Ankle Ability Measure (FAAM) Tool.
Time Frame: One year
Population: No participants randomized or treated.
Arm/Group | Bupivacaine Hydrochloride and Betamethasone Sodium Phosphate | Bupivacaine Hydrochloride
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: participant withdrew before randomization and prior to any assessment of adverse events.
Description: No participants treated on this trial therefore no adverse events were collected on the study.
Arm/Group | Bupivacaine Hydrochloride and Betamethasone Sodium Phosphate | Bupivacaine Hydrochloride
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes